CLINICAL TRIAL: NCT06909006
Title: Obesity and Semaglutide in Type 1 Diabetes Therapy: A Multicentre, Randomised, Double-Blinded, Placebo-Controlled, Investigator-Initiated Trial
Brief Title: Semaglutide Treatment in Type 1 Diabetes
Acronym: OBES1TY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Steno Diabetes Center Odense (Other); Zealand University Hospital (Other); Steno Diabetes Center Aarhus (SDCA), Aarhus University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1304-0713
Record Dates: First submitted 2025-03-17; First posted 2025-04-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: Obesity in Diabetes; Obesity/Therapy; Type 1 Diabetes Mellitus (T1DM); Insulin Sensitivity/Resistance; Semaglutide; Lipidomics; Metabolomics; Weight Loss; Glycemic Control for Diabetes Mellitus
Keywords: Semaglutide; Obesity; Type 1 Diabetes; Obese Type 1 Diabetics; Insulin sensitivity; Insulin resistance; Weight loss; GLP1-RA; GLP1; Wegovy
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 1; Insulin Resistance; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Randomised, double-blinded, placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Active Comparator): Subcutaneous injection through injector pen with the active comparator Semaglutide once a week in monthly increasing doses as given: 0.25mg - 0.5mg - 1.0mg - 1.7mg - 2.4mg
  Interventions: Drug: Semaglutide 2.4mg
- Semaglutide placebo (Placebo Comparator): Visually identical injector pen without the active comparator.
  Interventions: Drug: Semaglutide placebo

INTERVENTIONS:
Drug: Semaglutide 2.4mg — The active comparator of the intervention is s.c. Semaglutide injection once a week in increasing doses every month from 0.25 mg to 0.5 mg to 1.0 mg to 1.7 mg to 2.4 mg and the placebo comparator is s.c. injection with a visually identical and same label pen as described for the active comparator
  Other Names: Active semaglutide
  Arms: Semaglutide
Drug: Semaglutide placebo — Visually identical and same label as the active comparator intervention
  Other Names: Placebo semaglutide
  Arms: Semaglutide placebo

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of semaglutide on body weight, insulin dose requirements and improvements in glucose control and safety aspects in regards to risk of hypoglycemia and diabetic ketoacidosis for patients with established Type 1 Diabetes.

DETAILED DESCRIPTION:
This is a multicentre, randomised, double-blinded, placebo-controlled and investigator-initiated trial aimed to investigate the efficacy of semaglutide in patients with Type 1 Diabetes.

Patients from all included diabetes care centres will at routine visits be screened for eligibility for the trial and offered participation. If accepted, the patients will be randomised to one of two intervention arms and undergo a series of different examinations prior to start of the intervention.

The two arms consist of treatment with subcutaneous semaglutide injections or subcutaneous injections with semaglutide placebo. The baseline examinations entail documentation of insulin doses, dietary patterns, diabetes distress and treatment satisfaction questionnaires, anthropoimetric data (height, weight and calculation of BMI, waist circumference, waist-hip-ratio), blood work (HbA1c, fasting glucose, fasting c-peptide, lipids, liver and kidney markers incl. Fib-4-scoring, hematology, hsCRP), ECG, capturing of data from continuous/flash glucose monitors.

The first 40 included in the study from the centres of SDCA and NOH will further be examined through hyperinsulinemic euglycemic clamps to determine their insulin sensitivity and asses their transcriptome through muscle and fat cell biopsies in relation to the clamp and also be assessed through DXA scans to look at body composition and bone density.

Patients will then be handed out their trial drug-pens and start the uptitration proces.

The efficacy of semaglutide will be evaluated through the above mentioned array of different investigations by comparing parameters prior to trial drug start, during (throughout the study period), at the end of the drug and at a 6 week post-study followup in an intention-to-treat analysis primarily and secondarily a per-protocol analysis.

The safety will be assessed through evaluation of standardized adverse event reporting (including hypoglycemic events and diabetic ketoacidosis).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes for more than 3 years
* BMI ≥ 30 or ≥ 27 and atleast one comorbidity (hypertension, hypercholesterolemia, microalbuminuria, ischemic heart disease, history of stroke, atherosclerosis or arthrosis

Exclusion Criteria:

* Treated with GLP1-RAs within last 6 months
* Known intolerance for semaglutide
* Other forms of diabetes
* Pregnant or nursing women
* Fertile women not using chemical (hormonal) or mechanical (spiral) contraceptives
* Liver disease with elevated plasma alanine aminotransferase (ALT) > five times and plasma aspartate aminotransferase (AST) > five times the upper limit of normal (measured at visit 0 with the possibility of one repeat analysis within a week, and the last measured value as being conclusive)
* Acute or chronic pancreatitis
* Cancer, unless in complete remission for > 5 years or unless basocellular carcinomas
* History of thyroid adenoma or carcinoma
* Alcohol/drug abuse
* Other concomitant disease or treatment that according to the investigator's assessment makes the patient unsuitable for study participation
* Receipt of an investigational drug within 30 days prior to visit 0 / Simultaneous participation in any other clinical intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Body weight | 74 weeks
  Body weight will be measured both prior to and following treatment for 68 weeks with either semaglutide or placebo. Changes in body weight will be compared for the two intervention arms, before, throughout and at the end of treatment and then at followup 6 weeks later.

SECONDARY OUTCOMES:
Systolic blood pressure | 74 weeks
  Systolic blood pressure will be assessed at randomization and evaluated for changes throughout, at the end of treatment and at followup 6 weeks later.
Diastolic blood pressure | 74 weeks
  Diastolic blood pressure will be assessed at randomization and evaluated for changes throughout, at the end of treatment and at followup 6 weeks later.
Resting heart rate | 74 weeks
  Systolic blood pressure will be assessed at randomization and evaluated for changes throughout, at the end of treatment and at followup 6 weeks later.
Waist circumference | 74 weeks
  Waist circumference will be assessed and evaluated for changes during and after treatment for 68 weeks with semaglutide compared to before treatment.
Hip-waist-ratio | 74 weeks
  Hip-waist-ratio will be assessed and evaluated for changes during and after treatment for 68 weeks with semaglutide compared to before treatment.
Hemoglobin | 74 weeks
  Blood samples will be analyzed to assess hemoglobin before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Leucocytes | 74 weeks
  Blood samples will be analyzed to assess leucocytes levels before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Thrombocytes | 74 weeks
  Blood samples will be analyzed to assess thrombocytes levels before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
HbA1c | 74 weeks
  Blood samples will be analyzed to assess HbA1c before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Fasting plasma-glucose | 74 weeks
  Blood samples will be analyzed to assess fasting plasma-glucose before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Fasting c-peptide | 74 weeks
  Blood samples will be analyzed to assess fasting c-peptide before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Total cholesterol | 74 weeks
  Blood samples will be analyzed to assess total cholesterol before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
HDL cholesterol | 74
  Blood samples will be analyzed to assess HDL cholesterol before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
LDL cholesterol | 74 weeks
  Blood samples will be analyzed to assess LDL cholesterol before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
VLDL cholesterol | 74 weeks
  Blood samples will be analyzed to assess VLDL cholesterol before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Triglycerides | 74 weeks
  Blood samples will be analyzed to assess triglycerides levels before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
non-HDL cholesterol | 74 weeks
  Blood samples will be analyzed to assess non-HDL cholesterol before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Sodium | 74 weeks
  Blood samples will be analyzed to assess sodium before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Potassium | 74 weeks
  Blood samples will be analyzed to assess potassium before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Creatinine/eGFR | 74 weeks
  Blood samples will be analyzed to assess creatinine levels to calculate estimated Glomerular Filtration Rates (eGFR, based on sex, age and creatinine leve) before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Alanine transaminase (ALT) | 74 weeks
  Blood samples will be analyzed to assess alanine transaminase (ALT) before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Aspartate transaminase (AST) | 74 weeks
  Blood samples will be analyzed to assess aspartate transaminase (AST) before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Fibrosis-4-score (Fib-4) | 74 weeks
  Blood samples will be analyzed for fibrosis-4-scores (based on age, thrombocytes, ALT and AST) before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Amylase | 74 weeks
  Blood samples will be analyzed to assess pancreatic amylase before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Lipase | 74 weeks
  Blood samples will be analyzed to assess pancreatic lipase before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
High sensitivity C-reactive protein (hsCRP) | 74 weeks
  Blood samples will be analyzed to assess high sensitivity C-reactive protein (hsCRP) before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Albumin | 74 weeks
  Blood samples will be analyzed to assess serum albumin before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Ketones | 74 weeks
  Blood samples will be analyzed to assess total serum ketones before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up
CGM data - Time in range (TIR) | 68 weeks
  Data from CGMs will be analyzed to asses time in range (TIR) before treatment and evaluated for changes in TIR throughout the 68-week regimen and at its conclusion.
CGM data - Time in tight range (TITR) | 68 weeks
  Data from CGMs will be analyzed to asses time in tight range (TITR) before treatment and evaluated for changes in TITR throughout the 68-week regimen and at its conclusion.
CGM data - Time above range (TAR) | 68 weeks
  Data from CGMs will be analyzed to asses time above range (TAR) before treatment and evaluated for changes in TAR throughout the 68-week regimen and at its conclusion.
CGM data - Time below range (TBR) | 68 weeks
  Data from CGMs will be analyzed to asses time in range (TBR) before treatment and evaluated for changes in TBR throughout the 68-week regimen and at its conclusion.
CGM data - coefficient of variation (CV) | 68 weeks
  Data from CGMs will be analyzed to asses coefficient of variation (CV) before treatment and evaluated for changes in CV throughout the 68-week regimen and at its conclusion.
Total daily dose of insulin | 74 weeks
  Total daily dose will be assessed at randomization and evaluated for changes throughout treatment regimen, at the end of study and at six weeks followup through the use of insulin dose diaries.
Insulin sensitivity | 68 weeks
  For a subgroup consisting of the first 40 patients from two specified sites: Insulin sensitivity will be assessed through the golden standard hyperinsulinemic euglycemic clamping method. This will be done before treatment and at the end of treatment.
Fat percentage | 68 weeks
  For a subgroup consisting of the first 40 patients from two specified sites: The fat percentage is measured by DXA scan at randomisation and at end-of-treatment.
Lean mass | 68 weeks
  For a subgroup consisting of the first 40 patients from two specified sites: Lean body mass is measured by DXA scan at randomisation and at end-of-treatment.
Bone density (through bone mineral content) | 68 weeks
  For a subgroup consisting of the first 40 patients from two specified sites: Bone density (through bone mineral content) is measured by DXA scan at randomisation and at end-of-treatment.
Omics / Metabolome | 74 weeks
  For a subgroup consisting of the first 40 patients from two specified sites: Blood samples will be analyzed to assess metabolomic profile (entailing both lipidome and proteome) before treatment and evaluated for changes throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up
Muscle tissue biopsy | 68 weeks
  For a subgroup consisting of the first 40 patients from two specified sites: Muscle tissue biopsies will be taken to assess changes in transcriptome at randomisation and at end-of-treatment.
Fat tissue biopsy | 68 weeks
  For a subgroup consisting of the first 40 patients from two specified sites: Fat tissue biopsies will be taken to assess changes in transcriptome at randomisation and at end-of-treatment.
Electrocardiogram | 68 weeks
  Electrocardiograms (ECG) will be recorded at initiation and end of treatment period to assess and evaluate if any rhytm changes occur.

OTHER OUTCOMES:
Patient reported outcome measures - Dietary patterns | 74 weeks
  Questionnaires (DNBCs FFQ) will be analyzed to evaluate changes in dietary patterns before treatment, throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Patient reported outcome measures - Diabetes treatment satisfaction | 74 weeks
  Questionnaires (DTSQ-s and DTSQ-c) will be analyzed to evaluate changes in diabetes treatment satisfaction before treatment, throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Patient reported outcome measures - Diabetes distress | 74 weeks
  Questionnaires (PAID) will be analyzed to evaluate changes in diabetes treatment satisfaction before treatment, throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.
Adverse events | 74 weeks
  Tolerability will be assessed through standardized adverse event reporting (including episodes of hypoglycemia) throughout the 68-week regimen, at its conclusion, and again six weeks post-treatment during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F Dejgaard, MD, ph.d., endocrinologist, Study Chair — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request for it.
Supporting Information: Study Protocol, SAP, CSR